CLINICAL TRIAL: NCT03878901
Title: Establishment of Systemic Prevention and Management for Perioperative Hypothermia and Its Effect on Patients Outcome-a Prospective Multiple Centers Randomized Controlled Study
Brief Title: Systemic Prevention and Management for Perioperative Hypothermia and Its Effect on Patients Outcome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Xuanwu Hospital, Beijing (Other); Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, Jie YI, Vice director, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Hypothermia2018
Record Dates: First submitted 2019-03-13; First posted 2019-03-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Hypothermia; Anesthesia
Keywords: hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Sham Comparator): Cotton Blanket Warming (CBW) starts 30 min preoperatively and then continues throughout the entire operation.
  Interventions: Other: passive warming
- warm group (Experimental): Warm according to different hypothermia risk for low risk ---Forced-air warming(FAW) starts at least 30 min preoperatively and then Cotton Blanket Warming (CBW) continues throughout the entire operation.
  moderate risk---Forced-air warming(FAW) starts at least 30 min preoperatively and then Cotton Blanket Warming (CBW) and fluid warming continues throughout the entire operation.
  high risk ----Forced-air warming(FAW) starts at least 30 min preoperatively, FAW and fluid warming continues throughout the entire operation.
  Interventions: Combination Product: high risk warm; Combination Product: moderate risk warm; Combination Product: low risk warm

INTERVENTIONS:
Combination Product: high risk warm — Bair HuggerTM Forced-air Warming System to 30min pre- and entire operation warming, combined fluid warming
  Arms: warm group
Combination Product: moderate risk warm — 30 min prewarming The Bair HuggerTM Forced-air Warming System cotton blanket warming and fluid warming through operation
  Arms: warm group
Combination Product: low risk warm — 30 min prewarming The Bair HuggerTM Forced-air Warming System and cotton blanket warming through operation
  Arms: warm group
Other: passive warming — cotton blanket warming through operation
  Arms: control group

SUMMARY:
This is a randomized, single-blinded, multi-center study clinical trial to determine both clinical and health outcomes of stratified warm strategy to prevent intraoperative hypothermia. Participants enrolled into this trial will be from elective major surgery population in PUMC Hospital, Beijing Hospital and Xuanwu Hospital. investigators plan to enroll approximately 800 participants. Hypothermia risk will be evaluated through PREDICTOR model in all participants. According to hypothermia risk level, these participants will be stratefied into high, moderate and low risk group. Participants in each group will be randomly categorize into warm group and control group. Active warm and fluid warm strategy, prewarm and fluid warm strategy and only prewarm strategy are used for high risk, moderate risk and low risk patients seperately. For controll group traditional passive warm was used.

ELIGIBILITY:
Inclusion Criteria:

Age≥18 Core temperature preoperation ≥36.0 ℃ and ≤37.5℃ ASA I-III Informed consent

Exclusion Criteria:

* emergency operation
* uncontrolled diebete mellitus with insulin treatment （preoperative blood glucose>250mg/dL）
* hyperthyroidism and hypothyroidism
* Raynaud's disease
* patients with hematopathy and immune disease
* anticoagulant and non-steroid anti-inflammatory drug intake with 14 days before operation
* infectious fever within 4 weeks before operation
* laboratory abnomality as follow
* Hemoglobin≤10.0g/L
* Platelet≤100,000/ml
* White blood cell<3000/dl or>14,000/dl
* Fibrinogen<200mg/dL
* Thrombin time>40 second
* International normalized ratio<70%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of intraoperative hypothermia | During operation
  Core temperature<36℃

SECONDARY OUTCOMES:
The amount of Intraoperative blood loss/blood transfusion | During operation
Length of stay in PACU | Postoperative during in postanaesthesia care unit， up to 24 hours after surgery
The incidence of Surgical site infection | WIthin 30 days postoperative
Lenght of Stay in hospital | impatient period， up to 6 month after surgery
Lenght of Stay in ICU | impatient period， up to 6 month after surgery
Incidence of Adverse cardiovascular events | WIthin 6 month post operation
Incidence of shiver | during in postanaesthesia care unit， up to 24 hours after surgery
Mini-Mental State Examination (MMSE), | One day preoperation and 1 , 7，30 days postoperation
  It's a scare to evaluate cognitive function. Total score is 30 . Higher values represent a better cognitive function.
digit symbol substitution test | One day preoperation and 1 , 7，30 days postoperation
  The digit symbol substitution test is an evaluation tool used to assess cognitive functioning. It initially was part of the Wechsler Adult Intelligence Test (WAIS), a well-known test that measures an individual's attention. lower digit symbol test scores were correlated with a higher risk of developing dementia in both the five and 10 year groups.Higher values represent a better cognitive function.
Auditory Verbal Learning Test, | One day preoperation and 1 , 7，30 days postoperation
  a memory test that involves learning verbal material, usually single words presented in a list, that is continually presented over repeated trials. Higher values represent a better memory functions.
Color Word Stroop Test | One day preoperation and 1 , 7，30 days postoperation
  The Stroop Colour and Word Test (SCWT) is a neuropsychological test extensively used to assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute, well-known as the Stroop Effect. Higher values represent a better ability to inhibit cognitive interference.
digit span test. | One day preoperation and 1 , 7，30 days postoperation
  a memory test that involves remember a series of numbers test short time memory Higher values represent a better memory functions.
postoperative cognitive dysfunction incidence | One day preoperation and 1 , 7，30 days postoperation
  * Z score=（postoperative score-preoperative core）/SD of non-surgical group
  * Two or more than two item in cognitive examination Z score<-1.96
  * Z score=（postoperative score-preoperative core）/SD of non-surgical group Two or more than two item in cognitive examination Z score<-1.96

CONTACTS AND LOCATIONS:
Overall Officials: Yuguang Huang, doctor, Study Chair — Peking Union Medcial College Hospital

IPD SHARING:
Plan to Share IPD: Undecided
There is not a plan to make IPD available.

REFERENCES:
- [Background] Yi J, Xiang Z, Deng X, Fan T, Fu R, Geng W, Guo R, He N, Li C, Li L, Li M, Li T, Tian M, Wang G, Wang L, Wang T, Wu A, Wu D, Xue X, Xu M, Yang X, Yang Z, Yuan J, Zhao Q, Zhou G, Zuo M, Pan S, Zhan L, Yao M, Huang Y. Incidence of Inadvertent Intraoperative Hypothermia and Its Risk Factors in Patients Undergoing General Anesthesia in Beijing: A Prospective Regional Survey. PLoS One. 2015 Sep 11;10(9):e0136136. doi: 10.1371/journal.pone.0136136. eCollection 2015. PMID 26360773
- [Result] Yi J, Zhan L, Lei Y, Xu S, Si Y, Li S, Xia Z, Shi Y, Gu X, Yu J, Xu G, Gu E, Yu Y, Chen Y, Jia H, Wang Y, Wang X, Chai X, Jin X, Chen J, Xu M, Xiong J, Wang G, Lu K, Yu W, Lei W, Qin Z, Xiang J, Li L, Yao M, Huang Y. Establishment and Validation of a Prediction Equation to Estimate Risk of Intraoperative Hypothermia in Patients Receiving General Anesthesia. Sci Rep. 2017 Oct 24;7(1):13927. doi: 10.1038/s41598-017-12997-x. PMID 29066717
- [Result] Yi J, Lei Y, Xu S, Si Y, Li S, Xia Z, Shi Y, Gu X, Yu J, Xu G, Gu E, Yu Y, Chen Y, Jia H, Wang Y, Wang X, Chai X, Jin X, Chen J, Xu M, Xiong J, Wang G, Lu K, Yu W, Lei W, Qin Z, Xiang J, Li L, Xiang Z, Pan S, Zhan L, Qiu K, Yao M, Huang Y. Intraoperative hypothermia and its clinical outcomes in patients undergoing general anesthesia: National study in China. PLoS One. 2017 Jun 8;12(6):e0177221. doi: 10.1371/journal.pone.0177221. eCollection 2017. PMID 28594825

DOCUMENTS (2):
  • Informed Consent Form (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/01/NCT03878901/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/01/NCT03878901/Prot_SAP_001.pdf